CLINICAL TRIAL: NCT07238972
Title: Impact of Postoperative Intravenous Iron Supplementation on the Incidence of Long-term Anemia in Patients Undergoing Cardiac Surgery
Brief Title: Postoperative Intravenous Ferric Derisomaltose for Prevention of Long-term Anemia After Cardiac Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2025-1187
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Anemia; Iron Deficiencies; Iron Deficiency Anemia; Cardiac Surgery; Heart Valve Diseases
MeSH Terms: conditions — Anemia; Iron Deficiencies; Anemia, Iron-Deficiency; Heart Valve Diseases | interventions — ferric derisomaltose; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A parallel-arm, postoperative anemia treatment trial evaluating intravenous ferric derisomaltose versus placebo.
Who Masked: Participant
Masking Description: Double-blind; participants, care providers, investigators, and outcome assessors remain blinded until study completion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferric derisomaltose (Experimental): Participants receive a single intravenous dose of ferric derisomaltose 20 mg/kg (maximum 1,000 mg) diluted in 100 mL normal saline and infused over 30 minutes on postoperative day 1.
  Interventions: Drug: Ferric derisomaltose
- Placebo (Placebo Comparator): Participants receive an equal volume of 0.9% saline placebo via intravenous infusion over 30 minutes on postoperative day 1.
  Interventions: Drug: Placebo (0.9% saline)

INTERVENTIONS:
Drug: Ferric derisomaltose — Ferric derisomaltose is administered as a single intravenous infusion at 20 mg/kg (maximum 1,000 mg), diluted in 100 mL normal saline, infused over 30 minutes on postoperative day 1.
  Arms: Ferric derisomaltose
Drug: Placebo (0.9% saline) — The placebo consists of 100 mL of 0.9% normal saline administered intravenously over 30 minutes on postoperative day 1, matched in appearance and timing to the ferric derisomaltose infusion to maintain blinding.
  Arms: Placebo

SUMMARY:
Postoperative anemia is highly prevalent among patients undergoing cardiac surgery and is associated with delayed functional recovery, increased morbidity, and impaired long-term outcomes. Preoperative iron deficiency is common in this population and contributes to inadequate erythropoietic recovery after surgery. Functional iron deficiency frequently develops even in patients without preoperative deficiency due to blood loss, hemodilution, and inflammation-mediated disruption of iron homeostasis. Despite this clinical burden, standardized strategies for postoperative anemia management have not been established.

This prospective, randomized, double-blind, placebo-controlled clinical trial evaluates whether early postoperative intravenous iron supplementation improves long-term anemia outcomes in patients undergoing cardiac surgery with cardiopulmonary bypass. Adult patients with preoperative anemia (hemoglobin <13 g/dL) or iron deficiency (ferritin <100 ng/mL or transferrin saturation <20%) will be screened. Eligible participants with postoperative day (POD) 1 hemoglobin <10 g/dL will be randomized in a 1:1 ratio to receive either ferric derisomaltose (20 mg/kg, maximum 1,000 mg) or a matched placebo administered intravenously over 30 minutes on POD 1. All perioperative management outside the intervention follows current institutional standards.

The primary outcome is the incidence of anemia at 6 months following surgery. Secondary outcomes include perioperative hemoglobin trends, functional recovery assessed by cardiopulmonary exercise testing and the 6-minute walk test at 6 months, transfusion requirements, postoperative complications including MAKE-90 and STS major morbidity, and changes in biomarkers of erythropoiesis and iron metabolism (erythroferrone, erythropoietin, hepcidin, and iron profile). Blood samples for biomarker analysis are collected at predefined perioperative timepoints.

Ferric derisomaltose allows high-dose single-session iron repletion with a favorable safety profile and minimal risk of anaphylaxis when administered slowly. Prior studies in cardiac surgery and heart failure populations support its efficacy and safety at doses up to 20 mg/kg. The intervention is expected to facilitate erythropoietic recovery, reduce the duration of postoperative anemia, and improve long-term functional status. The trial aims to generate evidence to inform postoperative anemia management strategies in cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥19 years scheduled to undergo cardiac surgery requiring cardiopulmonary bypass Preoperative anemia defined as hemoglobin <13.0 g/dL, or preoperative iron deficiency defined as ferritin <100 ng/mL or transferrin saturation <20% Ability to understand the study information and provide written informed consent prior to surgery

Postoperative day 1 hemoglobin <10.0 g/dL on the first CBC following surgery (required for final enrollment)

Exclusion Criteria:

* Emergency surgery Preoperative major organ failure requiring intensive care unit management Active infection prior to surgery, including sepsis Active bleeding prior to surgery Pregnancy or breastfeeding Use of erythropoiesis-stimulating agents or intravenous iron therapy within 3 months prior to surgery Iron overload defined as ferritin ≥500 ng/mL or transferrin saturation ≥45% Aplastic anemia Hemolytic anemia Hemochromatosis or hemosiderosis Decompensated liver cirrhosis, acute hepatitis, or alcohol dependence Known hypersensitivity to intravenous iron formulations Participation in another clinical trial that may influence outcomes Inability to understand or provide informed consent due to language barriers, illiteracy, or cognitive impairment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Anemia at 6 Months After Cardiac Surgery | Postoperative 6 months
  Proportion of participants with anemia at 6 months following cardiac surgery, defined as hemoglobin <13.0 g/dL in males and <12.0 g/dL in females. Hemoglobin is assessed at routine outpatient follow-up using standard laboratory testing.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine Anesthesia and Pain Research Institute Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No